CLINICAL TRIAL: NCT04428892
Title: CLINICAL SIMULATION IN PHYSIOTHERAPY STUDENTS IN CLINICAL COMPETENCE FOR INTERACT WITH PEOPLE WITH LOW BACK PAIN. COLOMBIA
Brief Title: Simulation in Physical Therapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Collaborators: Facultad Ciencias de La Salud Universidad de Boyaca (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ENF-19-2017
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Simulation Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Simulation (Experimental): The group denominated SP received a teaching strategy based on a class session with simulated practice for decision-making in clinical skills when caring for a person with LBP. Each session lasted approximately 120 minutes, and the clinical case used for the SP sessions was subjected to face validity with experts in the area of study.
  Interventions: Behavioral: Pedagogyc Strategy
- Conventional Pedagogical strategy (Active Comparator): received a class session based on a "role playing" simulation strategy, structured for the same purpose established in the SP group. This session lasted approximately 120 minutes, and the learning environment was the classroom in which students assumed different roles to act out; some of them acted as people with LBP and others as physiotherapists
  Interventions: Behavioral: Pedagogyc Strategy

INTERVENTIONS:
Behavioral: Pedagogyc Strategy — Simulation can be used as a pedagogic tool that provides students with significant learning regarding decision-making in interacting with people, in this case patients with LBP. It is a potential strategy for developing diverse skills focused on the safety of the patient and the therapist.

SUMMARY:
This randomized trial included physiotherapy students, randomized in two groups, experimental one included simulation for developed competencies related to clinical reasoning in physiotherapy interventions for people with low back pain. The second group developed role-playing. this protocol allows us to compare two strategies with simulation for to promote clinical decisions in physiotherapy practice.

DETAILED DESCRIPTION:
Low back pain (LBP) is symptomatology with a high global prevalence; health professionals, including physiotherapists, must have the skills to create professional interaction plans that permit a better quality of life for consultants. Clinical simulation can be a pedagogic setting that facilitates students with adequate training to acquire skills that improve professional reasoning in this clinical situation. The objective of this study was to compare the effects of clinical simulation with a simulated patient (SP) versus simulation with role-playing (RP) in physiotherapy students for decision-making in clinical skills while caring for a person with LBP. Methods. An experimental study, with 42 participants from two Colombian universities, randomized into two groups (SP n = 21, RP n = 21). The clinical skill was evaluated during the interaction with a person with LBP for which the Objective Structured Clinical Examination (OSCE-ML) was validated for individuals with low back pain; thereafter, a pedagogical method was conducted that included clinical simulation and, finally, the OSCE-ML was applied again to compare both groups.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy students in five-semester from Universidad de La Sabana and Universidad de Boyacá

Exclusion Criteria:

* under-age subjects
* those who had been internally or externally transferred from another academic program in health,
* exchange students
* those repeating
* with prior experiences in simulated practice in other assignments

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
clinical reasoning | 1 Month
  The Objetive structured Clinical Evaluation (OSCE) was designed and validated, with the proposal to asses the physiotherapeutic clinical reasoning in Low Back Pain people, The OCSE have included 7 stations for assesing the clinical reasoning students.

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Sandoval, Tunja, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sandoval-Cuellar C, Alfonso-Mora ML, Castellanos-Garrido AL, Del Pilar Villarraga-Nieto A, Goyeneche-Ortegon RL, Acosta-Otalora ML, Del Pilar Castellanos-Vega R, Cobo-Mejia EA. Simulation in physiotherapy students for clinical decisions during interaction with people with low back pain: randomised controlled trial. BMC Med Educ. 2021 Jul 9;21(1):375. doi: 10.1186/s12909-021-02812-7. PMID 34243767